CLINICAL TRIAL: NCT03758859
Title: CLARITY Imaging Study: The Effect Of Cross-linked Sodium Hyaluronate On The Quality Of Optical Coherence Tomography Imaging
Brief Title: CLARITY Imaging Study
Acronym: CLARITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18SM4868
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Masking Description: Randomisation is between eyes i.e. eye exposed to blinking alone vs eye exposed to lubricant drops
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sodium hyaluronate eye drops (Experimental): the randomly allocated eye will receive sodium hyaluronate drops, followed by a repeat OCT scan; images are then evaluated for clarity by the masked assessor.
  Interventions: Other: sodium hyaluronate eyedrops

INTERVENTIONS:
Other: sodium hyaluronate eyedrops — sodium hyaluronate eyedrops administered - route ocular -topical

SUMMARY:
OCT image quality is necessary to provide accurate diagnostic information to ophthalmologists. The increasing resolution of imaging techniques will require ever more high standards of optical transmission through the cornea and tear film. Given that lubricant drops can improve optical transmission through the cornea, this study will attempt to quantify this. The primary objective is to assess the effect of cross-linked sodium hyaluronate on OCT image quality compared to the effect of blinking alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjectively deemed to have poor image quality by the photographer

Exclusion Criteria:

* Patients with a known adverse reaction to any of the constituents of the XLHA
* Patients wearing contact lenses
* Patients who have used eyedrops in the past 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Clarity of retinal images obtained by Optical Coherence Tomography. | immediately after the administration of drops.
  Signal strength of OCT scan

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yap, Principal Investigator — Imperial College NHS Trust
Locations (1):
- Western Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided